CLINICAL TRIAL: NCT01687803
Title: Evaluating the Health Benefits of Physical Activity Recommendations in the Dietary Guidelines
Acronym: FL52
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 200614442-2
Record Dates: First submitted 2012-09-11; First posted 2012-09-19 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Obesity; Sedentary Lifestyle; Body Weight
Keywords: Obesity; Sedentary lifestyle; Body weight; Physical fitness
MeSH Terms: conditions — Obesity; Sedentary Behavior; Body Weight | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical Activity (Experimental): Physical activity intervention will consist of brisk walking or other aerobic-type activities (6 days per week), resistance exercise (using free weights, resistance bands or weight stacks for weight lifting, 3 days per week), and 'active lifestyle' activities such as gardening, dancing, participation in sporting activities. The total time spent in these activities will add up to ~60 min/day for 6 days/week (~360 minutes per week).
  Interventions: Behavioral: Physical Activity
- Control (Other): The control group will maintain their usual level of physical activity and participate in testing protocols, record keeping, and interviews.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Physical Activity — Physical activity intervention that will consist of brisk walking or other aerobic-type activities (6 days per week), resistance exercise (using free weights, resistance bands or weight stacks for weight lifting, 3 days per week), and 'active lifestyle' activities such as gardening, dancing, participation in sporting activities. The total time spent in these activities will add up to ~60 min/day for 6 days/week (~360 minutes per week).
  Arms: Physical Activity
Behavioral: Control — The control group will maintain their usual level of physical activity and participate in testing protocols, record keeping, and interviews.
  Arms: Control

SUMMARY:
The overall goal of this study is to determine the health benefits associated with the 2005 Dietary Guidelines physical activity prescription in healthy, peri-menopausal women. The 2005 Dietary Guidelines specifically state that to avoid unhealthy weight gain, adults should participate in 60 minutes of moderate to vigorous intensity physical activity on most days of the week.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial conducted over a 6 to 7 month period. Subjects will be enrolled by cohorts and randomly assigned to one of two groups.

* Group 1 (PA): physical activity intervention that will consist of brisk walking or other aerobic-type activities (6 days per week), resistance exercise (using free weights, resistance bands or weight stacks for weight lifting, 3 days per week), and 'active lifestyle' activities such as gardening, dancing, participation in sporting activities. The total time spent in these activities will add up to ~60 min/day for 6 days/week (~360 minutes per week).
* Group 2 (CON): control group will maintain their usual level of physical activity and participate in testing protocols, record keeping, and interviews on the same schedule as PA. This group will be offered an opportunity to have a gym membership/access to the training facility after completion of the 6-month period of serving as controls.

The specific aims of this pilot study are to:

* Assess each participant's level of compliance/adherence
* Assess the dietary habits of study participants as they become more physically active.
* Identify barriers to physical activity in this specific population.
* Measure changes in body composition, physical fitness and energy expenditure.
* Evaluate changes in chronic disease risk factors.
* Determine if regular physical activity reduces chronic stress.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index: 18.5 to 29.9 kg/m2
* Peri-menopause, as determined by self-report of menstrual history and symptoms for previous 12 months
* Sedentary lifestyle

Exclusion Criteria:

* Individuals who are already physically active
* Pregnant or nursing within the last 6 months
* Plan to become pregnant during the study
* Musculoskeletal disease or disorder which is expected to limit participation in physical activity
* Orthopedic injuries
* Inflammatory arthritis or autoimmune disorders
* Neuromuscular disorders including multiple sclerosis, amyotrophic lateral sclerosis, Parkinson's disease
* Menopause confirmed
* Use of tobacco products
* Family history of premature cardiovascular disease as defined by the ACSM guidelines
* Cardiovascular including a history of cardiac arrest; coronary heart disease, complex ventricular arrhythmia or atrial arrhythmia at rest or with exercise, congestive heart failure, cardiomyopathy, hemodynamically significant valvular heart disease, left bundle block, cardiac pacemaker; implanted cardiac defibrillator; history of aortic aneurysm of at least 7 cm in diameter or aortic aneurysm repair; resting heart rate < 45 beats per minute or > 100 beats per minute
* Chronic lung disease resulting in dyspnea at rest or with minimal exertion, lung disease resulting in hypoxia or hypercapnia at rest or with exercise, pulmonary embolus within 6 months, active tuberculosis
* Presence of risk factors for cardiovascular or metabolic disease:
* Hypertension (SBP ≥140 mm Hg and/or DBP ≥ 90 mm Hg); hypertension treated by beta adrenergic blockers regardless of blood pressure
* Elevated fasting LDL cholesterol (≥160 mg/dL)
* Elevated fasting triglycerides (≥300 mg/dL)
* Diagnosed diabetes mellitus or elevated fasting glucose (≥126 mg/dL), adrenal disease, acromegaly, or thyroid disease requiring medication change or other treatment within the previous 3 months
* Weight change greater than 10 lbs in the preceding 6 months
* Medications: chronic corticosteroid use or need for oral corticosteroids more than twice in the last 12 months, antipsychotic medications, beta adrenergic blockers, medications for weight loss (including sibutramine, orlistat, phentermine, phendimetrazine, topiramate, zonisamide), immunosuppressants, amphetamines and other stimulants, and other medications known to influence body weight
* Travel plans that do not permit full participation

Ages: 42 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2006-10; Primary Completion 2009-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Change in compliance with exercise | 0, 3 and 6 months
  The Actiheart (MiniMitter, Bend OR) physical activity and heart rate logger is a motion sensor and heart rate monitor worn by subjects 24 hours per day(excluding bathing and swimming) for one week to determine the level of physical activity. Subjects will also use a pedometer to record the number of steps taken during their walking sessions. The Stanford 7 day Physical Activity recall questionnaire will also be used to assess physical activity.

SECONDARY OUTCOMES:
Change in dietary intake | 0, 6 months
  The 24-hour dietary recall will be used to assess usual dietary intake. Four recalls will be collected on non-consecutive days during the first and sixth months of the study. Additionally, the Healthy Eating Index for diet quality will be used to score the diets of subjects.
Change in body composition | 0, 3, and 6 months
  Body Composition is measured by dual energy x-ray absorptiometry (DEXA) using a whole body scan.
Change in Chronic Disease Risk Assessment | 0, 3 and 6 months
  Chronic Disease Risk Assessment includes blood pressure, fasting blood cholesterol, HDL cholesterol, LDL cholesterol, triacylglycerides, non-esterified fatty acids, ApoAI, ApoAII, and ApoB, glucose, insulin. Insulin sensitivity will be assessed by the homeostatic model utilizing fasting insulin and glucose values (fasting plasma insulin (mU/ml) X fasting plasma glucose (mmol/L)/22.5). High sensitivity C-Reactive Protein, inflammatory cytokines including IL-6 and TNF-α, Oxylipins and other markers of oxidative stress such as oxygen radical absorptive capacity will be analyzed in plasma samples.
Change in measures of stress | 0, 3 and 6 months
  At baseline and after three and six months of the exercise intervention participants will be asked to collect saliva samples for the assessment of salivary cortisol.
Change in aerobic fitness | 0, 3, and 6 months
  Maximal aerobic capacity is measured using a walking graded treadmill test. Indirect calorimetry will be used to measure oxygen consumption and carbon dioxide production continuously during the exercise test.
Change in measures of muscle strength | 0, 3, and 6 months
  Peak strength and muscle endurance of the musculature of the knee and shoulder will be measured using an isokinetic dynamometer. A measure of the maximum weight that can be moved for a single repetition (1-RM) will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy L Keim, PhD, Principal Investigator — USDA, ARS, Western Human Nutrition Research Center

REFERENCES:
- See also: USDA Western Human Nutrition Research Center — http://www.ars.usda.gov/Main/docs.htm?docid=11240